CLINICAL TRIAL: NCT03367065
Title: Dynamic Contrast Enhancement Computed Tomography Based Technic to Assess Gastro Intestinal Wall Perfusion : Feasibility Study
Acronym: PERFE-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PERFE-CT
Record Dates: First submitted 2016-08-26; First posted 2017-12-08 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Mesenteric Ischemia; Permeability CT Technics
MeSH Terms: conditions — Mesenteric Ischemia

ARMS (1):
- Dynamic contrast enhanced computerised tomography (Experimental)
  Interventions: Radiation: Dynamic contrast enhanced computerised tomography

INTERVENTIONS:
Radiation: Dynamic contrast enhanced computerised tomography

SUMMARY:
This feasibility study has therefore several aims:

1. construct a dedicated CT perfusion protocol for GIT wall perfusion;
2. used a two-compartment pharmacokinetic model which is more adapted that a unique compartment model;
3. from the image acquired, evaluate current parameters of perfusion including the permeability ones

ELIGIBILITY:
Inclusion Criteria:

* all patients over fifty years old with clinico-biological suspicion for acute GITischemia admitted at our institution

Exclusion Criteria:

* contra-indication to contrast agent injection as so defined by the European Society of UroRadiology in 2014
* inability to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
number of computerised tomography with interpretable data | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume HERPE, MD, Principal Investigator — CHU Poitiers
Locations (1):
- Chu Poitiers, Poitiers, Aquitaine, France